CLINICAL TRIAL: NCT00580242
Title: A Phase I Dose Escalating Study of Bortezomib and Lenalidomide in Patients With Untreated or Previously Treated, Primary and Secondary Non 5q- Del Myelodysplasia
Brief Title: A Phase 1 Dose Escalating Trial of Bortezomib in Combination With Lenalidomide in Patients With Myelodysplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene Corporation (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Karen Ballen, Director, Leukemia Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-006; RV-MDS-PI-0161
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Myelodysplasia
Keywords: Myelodysplasia
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts | interventions — Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This is a Phase I dose escalation trial with three cohorts of 3-6 patients each plus 10 additional patients (up to a maximum total of 28 patients) treated at the candidate maximum tolerated dose.Cohorts will receive increasing doses of bortezomib at 0.7, 1, and 1.3 mg/m2 on days 1, 4, 8, and 11 in combination with lenalidomide at 10 mg a day for Days 1-21. Each cycle will be 28 days. Patients will receive up to 9 cycles of treatment, with efficacy assessed after 3, 6, and 9 cycles.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — First cohort: Bortezomib 0.7mg/m2 IV on Days on Days 1, 4, 8, and 11. Patients may receive up to 9 cycles with each cycle lasting a total of 28 days
  Other Names: Velcade
Drug: Bortezomib — Second cohort: Bortezomib 1mg/m2 IV on Days 1, 4, 8, and 11 Patients may receive up to 9 cycles with each cycle lasting a total of 28 days
  Other Names: Velcade
Drug: Bortezomib — Third Cohort: Bortezomib 1.3mg/m2 IV on Days 1, 4, 8, and 11 of each cycle Patients may receive up to 9 cycles with each cycle lasting a total of 28 days
  Other Names: Velcade
Drug: Lenalidomide — Lenalidomide 10 mg PO QD on Days 1 -21 followed by a 7 day rest period
  Other Names: Revlimid

SUMMARY:
This study proposes using bortezomib in cohorts of 3-6 patients at the doses of 0.7, 1, and 1.3 mg/m2 on days 1, 4, 8, and 11 to determine the MTD in combination with lenalidomide 10 mg a day, for 21 days of a 28 day treatment cycle for patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
Currently, there are no curative therapies for myelodysplasia except for allogeneic stem cell transplantation. Both lenalidomide and bortezomib have activity as single agents in patients with myelodysplasia. This study proposes using bortezomib in cohorts of 3-6 patients at the doses of 0.7, 1, and 1.3 mg/m2 on days 1, 4, 8, and 11 to determine the MTD in combination withlenalidomide 10 mg a day, for 21 days of a 28 day treatment cycle. The planned bortezomib doses have been evaluated in previous Phase I clinical studies in similar patient populations and have been safe and well tolerated in a twice-weekly schedule of administration. Lenalidomide has been shown to have efficacy in myelodysplasia. The combination of lenalidomide and bortezomib has been used in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be untreated or previously treated.
* Age > 18 years
* Able to adhere to study schedule and other protocol requirements
* Unequivocal clinicopathologic diagnosis of myelodysplastic syndrome, non 5q- deletion.
* Patients may have had prior chemotherapy or radiotherapy for another malignancy or myelodysplasia as long as it was completed at least 4 weeks (6 weeks for nitrosureas) prior to initiation of therapy.
* ECOG performance status of 0-2 (Appendix 10.3)
* Life expectancy greater than 3 months
* Total bilirubin ≤ 2.0 mg/dl, ALT and AST ≤ 3 X the upper limit of normal (ULN), creatinine < 2.0 mg/dl all within 28 days prior to enrollment.
* Patients must give voluntary written informed consent and HIPAA authorization before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Absolute neutrophil count > 0.5 x 10 (9)/l
* Platelet count > 30 x 10 (9)/l
* Prior treatment with 5-azacytidine is encouraged, but not required.
* Patients may have had prior treatment for MDS, including single agent lenalidomide or bortezomib.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50mIU/ml within 10-14 days prior to and within 24 hours of prescribing lenalidomide and must commit to abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control,at least 4 weeks before starting taking lenalidomide. FCBP must agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.
* All study participants must be registered into the mandatory RevAssist Program®, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

* Ejection fraction < 40%
* Patients who have had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the consent form.
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with major surgery within the 28 days prior to trial enrollment.
* Patients with ≥ Grade 2 peripheral neuropathy or active herpes infection
* Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cirrhosis, chronic obstructive or restrictive pulmonary disease, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrythmia.
* Patients with secondary MDS that require concurrent therapy for the primary cancer diagnosis.
* The development of erythema nodosum as characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patient with hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. . Lactating females must agree not to breast feed while taking lenalidomide.
* Patient has received an investigational drug within 28 days of enrollment.
* Known hypersensitivity to thalidomide or lenalidomide
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Establish the maximally tolerated dose of bortezomib, up to 1.3 mg/m2/day, that can be administered in combination with lenalidomide in patients with primary and secondary non 5q del myelodysplasia who are untreated or previously treated. | 3, 6 and 9 months

SECONDARY OUTCOMES:
Assess efficacy in terms of the number of patients experiencing a decrease in blast percentage | 3, 6 and 9 months
Assess efficacy in terms of the number of patients experiencing a decrease in transfusion requirements | 3, 6 and 9 months
Determine the toxicity profile of bortezomib when used in combination with lenalidomide for patients with myelodysplasia | 3, 6 and 9 months
Determine the time (days) to transfusion independence | 3, 6 and 9 months
Determine the duration of response | 3, 6 and 9 months
Determine if molecular markers can predict responsiveness to treatment (for consenting patients) | 3, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts